CLINICAL TRIAL: NCT03228784
Title: The Effect of Ablation Depth on Dry Eye After LASIK Treatment of Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosny Ahmed Zein, Principle Investigator, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5780
Record Dates: First submitted 2017-07-14; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Incidence and Severity of Dry Eye After Myopic LASIK
MeSH Terms: interventions — Keratomileusis, Laser In Situ

INTERVENTIONS:
Procedure: LASIK
  Other Names: Corneal Flap creation with mechanical microkeratome and stromal ablation with Excimerr laser.

SUMMARY:
The study tried to find the relation between ablation depth and degree of dryness after LASIK treatment of myopic patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 21 years
* Normal Pentacam maps
* Myopia with spherical equation less than 12 D
* Corneal thickness ≥ 500 Microns
* Calculated residual stromal bed ≥ 280 microns
* No signs or symptoms of dry eye.

Exclusion Criteria :

* Keratoconus and forme fruste keratoconus
* Auto-immune diseases
* History of dry eye or previous use of tear substitutes
* Previous ocular surgery
* Pregnant or lactating women.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2014-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dry eye | 6 months
  Schirmer 1 test in millimeters
Degree of dryness | 6 months
  Tear break up time in seconds

IPD SHARING:
Plan to Share IPD: No